CLINICAL TRIAL: NCT01433562
Title: Combination of DLBS1425 With Anthracyclin-based Regimen as a Neoadjuvant Therapy in Subjects With Stage II or III Breast Cancer
Brief Title: Efficacy and Safety of DLBS1425 as Neoadjuvant in Stage II or III Breast Cancer Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Dexa Medica Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DLBS1425-0310
Record Dates: First submitted 2011-09-09; First posted 2011-09-14 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2013-05

CONDITIONS: Breast Cancer
Keywords: breast cancer; neoadjuvant therapy; Stage II/III
MeSH Terms: conditions — Breast Neoplasms | interventions — DLBS 1425

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DLBS1425 (Experimental)
  Interventions: Drug: DLBS1425
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo DLBS1425

INTERVENTIONS:
Drug: DLBS1425 — DLBS1425 capsule 150 mg thrice daily for 3 cycles @ 21 days. CAF (Cyclophosphamide (500 mg/m2 iv), Doxorubicin 50 mg/m2 iv, Fluorouracil 500 mg/m2 iv) or CEF (Cyclophosphamide 500 mg/m2 iv, Epirubicin 70 mg/m2 iv, Fluorouracil 500 mg/m2 iv) regimens on Day-1 of every cycle for the total of 3 cycles.
  Arms: DLBS1425
Drug: Placebo DLBS1425 — Placebo DLBS1425 capsule thrice daily for 3 cycles @ 21 days. CAF (Cyclophosphamide (500 mg/m2 iv), Doxorubicin 50 mg/m2 iv, Fluorouracil 500 mg/m2 iv) or CEF (Cyclophosphamide 500 mg/m2 iv, Epirubicin 70 mg/m2 iv, Fluorouracil 500 mg/m2 iv) regimens on Day-1 of every cycle for the total of 3 cycles.
  Arms: Placebo

SUMMARY:
This is a 2-arm, randomized, double-blind, placebo-controlled study aiming to determine the efficacy and safety of DLBS1425 in combination with anthracyclin-based regimen as a neoadjuvant therapy in subjects with previously untreated stage II or III (operable) breast cancer.

The anthracyclin-based regimen in the study will be either CAF/iv and CEF/iv only. The neoadjuvant anthracyclin-based chemotherapy will be given for 3 cycles. The length of each cycle will be 21-28 days.

DETAILED DESCRIPTION:
The duration of treatment for each subject will be 63 - 84 days (or 3 cycles). The cycle will be initiated at Day-1 (D1 of the 1st cycle). The subsequent cycles will start on Day-22 (D1 of the 2nd cycle) and Day-43 (D1 of the 3rd cycle). DLBS1425 capsules will be administered orally every day (starting from D1 of each cycle) during the study period. All subjects will be under direct supervision of a medical doctor during the study period.

Clinical and laboratory examinations to evaluate investigational drug's efficacy and safety will be performed at baseline and at the end of every cycle over the study course; whilst breast-CT scan will be performed at baseline and at the end of study course.

In addition, at the end of study, at the discretion of Investigator and subjects' own willingness, subjects with good response to treatment (i.e. RECIST and pathological evaluation are regarded as complete or partial response) may continue their breast-cancer therapy with DLBS1425.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed stage II or III (operable) primary breast cancer
* Having radiologically evaluable and measurable lesion(s) of the primary tumor
* Karnofsky performance status 80 %
* Normal cardiac function: LVEF > 50 %
* Adequate hematological function: Hb ≥ 10.0 g/dL, WBC ≥ 3,000/mm3, ANC ≥ 1,500 /mm3, platelet count ≥ 100,000/mm3
* Adequate liver function: ALT ≤ 2.5 times upper limit of normal, total bilirubin level ≤ 1.5 times upper limit of normal
* Adequate renal function: serum creatinine ≤ 1.5 times upper limit of normal
* Able to take oral medication

Exclusion Criteria:

* Pregnancy or breast feeding subjects
* History of previous breast cancer (recurrent breast cancer)
* History of other cancer within the past 5 years
* Prior systemic treatment for the current breast cancer
* Prior preoperative topical treatments for the current breast cancer
* Uncontrolled or serious CVD
* Known or suspected hypersensitivity to any of the chemotherapeutic agents used in the study
* Any other serious disease state or medical condition which judged by investigator could interfere with trial participation or trial evaluation
* Concurrent herbal (alternative) medicines or food supplements suspected to have effect on breast cancer disease within 14 days prior to screening
* Severe psychological or neurological disorder or dementia that would preclude understanding of the informed consent
* Participation in any other clinical studies within 30 days prior to screening

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Clinical response as measured by RECIST | 63 - 84 days
  Best overall response rate defined as proportion of subjects with either complete or partial response, according to the RECIST criteria at the end of study.

SECONDARY OUTCOMES:
Rate of clinical response | 21 - 84 days
  Rate of clinical response categorized as complete response, partial response, stable, and progressive disease, which will be evaluated clinically at the end of every cycle
Rate of pathological complete response (after surgery) | 7 - 14 days after the last cycle
  Pathological complete response based on histological examination will be assessed after surgery. The surgery itself will be performed within 7 - 14 days after the last cycle.
Rate of potential breast-conserving procedure | 63-84 days
  Rate of potential breast-conserving procedure as assessed by mammography, will be evaluated at the end of study.
The change level of relevant biomarkers | 21 - 84 days
  Relevant biomarkers related to breast cancer (CEA, CA-15.3, and serum LDH)will be measured at baseline and at the end of every cycle.
Haematology | 21-84 days
  Haematology parameters (Haemoglobin level, Haematocrit, red blood cell count, white blood cell count as well as its differentials, and platelet count) will be evaluated at baseline and the end of every cycle.
Liver Function | 21-84 days
  Liver function parameters (alkaline phosphatase, ALT, AST, bilirubin levels)will be measured at baseline, and the end of every cycle.
Renal Function | 21-84 days
  Renal Function (serum creatinine and Blood urea nitrogen levels) will be measured at baseline and the end of every cycle.
Cardiac function | 63-84 days
  Cardiac function will be assessed by ECHOcardiography at baseline and the end of study.
Adverse Events | 1 - 84 days
  Adverse events as well as number of subjects experienced the events will be observed and evaluated during the study period (from the first dose of study medication taken (Day 1) till the end of study treatment (Day 63 - Day 84).
The improvement of quality of life | 21 - 84 days
  The improvement of quality of life of the subjects as measured at baseline and at the end of each treatment cycle, using Functional Assessment of Cancer Therapy-General (FACT-G) Questionnaire (FACIT.org)

CONTACTS AND LOCATIONS:
Overall Officials: Heru Purwanto, MD, SpB(K)Onk, MSc., Principal Investigator — Surgery-Oncology Division, Department of Surgery, Faculty of Medicine, University of Airlangga / Dr. Soetomo Hospital
Locations (1):
- Surgery-Oncology Division, Department of Surgery, Faculty of Medicine, University of Airlangga / Dr. Soetomo Hospital, Surabaya, East Java, Indonesia